CLINICAL TRIAL: NCT07167277
Title: Impact of Whey Protein on Frailty - a Pilot Study
Brief Title: The Impact of Whey Protein on Frailty in Older Adults Classified as Pre-frail
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00161162
Record Dates: First submitted 2025-08-11; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pre-frail; Pre-Frail Older Adults; Cognition; Physical Function; Dietary Intake Assessment; MRI
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey Protein (Experimental): Participants will receive the dietary intervention. Participants will take one serving of whey protein per day.
  Interventions: Dietary Supplement: Whey Protein
- Placebo (Active Comparator): Participants will receive a placebo. Participants will take one serving of placebo per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Whey Protein — 24g of whey protein will be given to the participant to be consumed daily. Participants will be asked to consume 1 serving per day for 3 months.
  Arms: Whey Protein
Dietary Supplement: Placebo — A calorie matched serving of carbohydrate powder will be given to participants to consume daily. Participants will be asked to consume 1 serving per day for 3 months.
  Arms: Placebo

SUMMARY:
This pilot study aims to determine the impact of whey protein supplementation on brain antioxidant levels and to assess the effects of whey protein supplementation on physical function, body composition, and cognition in pre-frail older adults.

DETAILED DESCRIPTION:
Frailty is characterized by weakness, muscle loss, and physical impairment. It is suggested that long term oxidative stress might contribute to frailty. Glutathione (GSH), an antioxidant in cells, is needed to combat oxidative stress. Whey protein has the potential to increase brain antioxidant (GSH) levels by aiding in antioxidant synthesis. Frail older adults under-consume protein compared to healthy older adults.

Researchers want to see if supplementing with whey protein will improve brain antioxidant status in pre-frail older adults. They will measure this by using special Magnetic Resonance Imaging (MRI) scans.

Participants will be asked to complete a total of 4 study visits, all taking place on the University of Kansas Medical Center (KUMC) main campus. Two of these visits will include an MRI scan. Participation will last about 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Pre-frail according to Fried's phenotype
* Age 65 to 85
* Speak English as primary language and able to read and write in English
* Stable medication for ≥ 30 days
* Not already taking whey protein over the past 30 days

Exclusion Criteria:

* Acute or chronic kidney disease
* Recent major health concerns
* Insulin-requiring diabetes
* Cancer requiring chemotherapy or radiation within the past 5 years
* Cardiac event (i.e., MI, etc.) in the past year
* Dementia or neurodegenerative disease
* Clinical trial or investigational drug or therapy participation within 30 days of the screening visit or during enrollment in the current study
* MRI contraindications (pacemaker, aneurysm clips, artificial heart valves, metal fragments, foreign objects or claustrophobia)
* Dairy Allergy or excluding dairy from diet for other reasons
* Weight > 350 lbs.
* The presence of major psychiatric disorders within the past 3 years including depression, anxiety, and alcohol (over 3 drinks/day or a total of 18 drinks/week) or drug abuse.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in brain glutathione (GSH) levels measured using MRI scans. | Changes from baseline to 3 months.
  Brain GSH levels will be measured using 3T MRI scans.

SECONDARY OUTCOMES:
Assess the change in physical function by measuring balance resistance, sit-to-stand, muscle strength and performance. | Changes from baseline to 3 months.
  Balance resistance will be measured with a pressure-sensitive walkway. Sit-to-stand will be measured by number of repetitions in 30 seconds and the time to complete 5 repetitions. Muscle strength and performance will be measured by grip strength and gait speed. Grip strength is measured 3 times and averaged. Gait speed is measured with a 15-foot walk test and will be measured twice.
Assess body composition with a bioelectrical impedance analysis (BIA) device. | Changes from baseline to 3 months.
  To measure, subjects will stand on the device, covering the electrodes with their hands and feet. The measure takes less than 2 minutes.
Assess cognition using the NIH Toolbox cognition battery. | Changes from baseline to 3 months.
  The NIH Toolbox cognition battery will include 5 tests resulting in a composite score. The exam will be administered on an iPad device.

CONTACTS AND LOCATIONS:
Overall Officials: Debra K Sullivan, Principal Investigator — Department of Dietetics and Nutrition
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No